CLINICAL TRIAL: NCT06360809
Title: Prehabilitation Exercise Program in Breast Cancer: Effects on Quality of Life and Tumor Microenvironment (PEP_BC)
Acronym: PEP_BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Nacional d'Educacio Fisica de Catalunya (Other)
Collaborators: ICFO - The Institute of Photonics Sciences (Unknown); Hospital Clinic of Barcelona (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Albert Busquets Faciaben, Principal Investigator, Institut Nacional d'Educacio Fisica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024 PARINEFC 00001
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical exercise; tumor microenvironment; oxidative hemodynamics; near-infrared spectroscopy; diffuse correlation optical spectroscopy; prehabilitation therapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP group (Experimental): Breast cancer patients involved in a prehabilitation physical exercise program
  Interventions: Behavioral: Prehabilitation exercise program
- CON group (No Intervention): Breast cancer patients not involved in a prehabilitation physical exercise program

INTERVENTIONS:
Behavioral: Prehabilitation exercise program — After the allocation, the intervention will consist of a prehabilitation program lasting 4 weeks. Each week, there will be three sessions, with one being face-to-face and the other two being unsupervised sessions but with online video-support. Face-to-face sessions will be organized in small groups, and each patient of the PEP group will have an individualized plan based on data obtained during the initial assessment. Each session will include a combination of strength training and moderate aerobic training in a circuit format with movements especially involving the upper body.
  Arms: PEP group

SUMMARY:
To improve the health and quality of life of breast cancer (BC) patients, researchers are focusing on prehabilitation strategies like physical exercise, preparing patients both mentally and physically for clinical and surgical procedures, potentially reducing complications. Physical exercise is also recognized as pivotal in optimizing chemotherapy. It can improve blood flow and oxygen supply in the microenvironment of the tumor (MT), potentially enhancing chemotherapy effectiveness. Although previous research has shown the benefits of preoperative exercise combined with chemotherapy in various cancer types, including BC, further investigation is needed into the exact effects of prehabilitation exercise (PE) on MT physiology.

This study aims to provide valuable insights into the potential benefits of PE for BC patients and its impact on the tumor microenvironment. The hypothesis is that PE in BC patients will improve their quality of life, reduce fatigue, increase muscle mass, decrease fat mass, and enhance physical fitness. Additionally, beneficial acute hemodynamic changes, particularly increased blood flow following PE sessions, and hemodynamic adaptations involving higher levels of oxygenated hemoglobin, increased blood flow, greater oxygen saturation, and a higher metabolic rate of oxygen, are expected.

The study will include 76 participants aged 18-65 years, meeting specific criteria such as a diagnosis of hormone receptor-positive BC, no medical contraindications for exercise, no metastatic cancer, and no structured exercise in the last six months. These participants will be randomly assigned to a PE group or a control group. The study will consist of three phases: Phase 1 involves pre-intervention assessments, Phase 2 includes a 4-week PE intervention with three weekly sessions, and Phase 3 encompasses post-intervention and post-surgery assessments. The 4-week PE intervention in Phase 2 will include strength and aerobic training. Quality of life and fatigue assessments will use questionnaires, and measurements will be made for fat mass, lean mass, bone density, and cardiorespiratory fitness. Strength measurements will be taken, and shoulder mobility will be evaluated. Hemodynamics of the MT will be assessed using a hybrid device combining Near-Infrared Spectroscopy and Diffuse Correlation Spectroscopy with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18 and 65 years.
* Have a diagnosis of hormone receptor-positive breast cancer (ER and PR).
* Have no medical contraindications that prevent them from participating in physical exercise.
* Have four weeks period between diagnosis and surgery

Exclusion Criteria:

* Being diagnosed of another primary and/or secondary tumor or being in metastatic stage.
* Presence of uncontrolled serious medical illness
* Presence of any medical, psychological or social problem that could seriously interfere with the patient's participation in the study
* Those who have engaged in structured physical exercise in the last 6 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life score | 0, 28,and 35 days
  Quality of life will be assessed using the 'European Organisation for Research and Treatment of Cancer Quality ofLife Questionnaire' (EORTC QLQ-C30). This questionnaire has three different scales: (1) Global health status with 2 items scored from 1 to 7, (2) Functional scales with 15 items scored from 1 to 4, and (3) Symptom scales with 13 items scored from 1 to 4. All of the raw scores from the scales are transformed to values from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a healthy level of functioning, a high score for the global health status represents a high quality of life, but a high score for a symptom scale represents a high level of symptomatology.
Cancer quality of life score | 0, 28,and 35 days
  Cancer quality of life will be assessed using the 'European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer' (EORTC QLQ-BR23). This questionnaire has two different scales: (1) Symptoms scale with 15 items scored from 1 to 4, and (2) Functional scales with 8 items scored from 1 to 4. All of the raw scores from the scales are transformed to values from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a healthy level of functioning, a high score for the global health status represents a high quality of life, but a high score for a symptom scale represents a high level of symptomatology.
Cancer-related fatigue | 0, 28,and 35 days
  For cancer-related fatigue evaluation, 'The Functional Assessment of Cancer Therapy - Breast' (FACT-B) will be administered.
Body composition | 0, 28,and 35 days
  To measure fat mass and lean mass (in absolute values, kg, or relative valeus. %) the dual X-ray absorptiometry (DEXA) technique will be used.
Bone density | 0, 28,and 35 days
  To measure the bone density (g/cm^2 or T score), the dual X-ray absorptiometry (DEXA) technique will be used.
Cardiorespiratory fitness | 0, 28,and 35 days
  Maximal oxygen volume (VO2 max) determine from an incremental test that will be conducted on a cycle ergometer with a portable gas analyzer to measure oxygen consumption.
Maximum isometric manual grip strength | 0, 28,and 35 days
  Maximum isometric manual grip strength measured using a handgrip dynamometer.
Upper body maximum strength | 0, 28,and 35 days
  Upper body tests involve pushing a fixed barbell with arms parallel to the ground and elbows at 90º similarly to a bench press. A force sensor will record force exerted during the strength tests.
Lower body maximum strength | 0, 28,and 35 days
  Lower body tests include performing knee extensions from a seated position with the knee at 90º against an immovable piece. A force sensor will record force exerted during the strength tests.
Shoulder range of motion | 0, 28,and 35 days
  Mobility will be measured using inertial sensors (gyroscope from a mobile) and a custom-made software to assess the maximum angle of motion (in degrees) in the three plans of motion.
Relative oxyhemoglobin concentration ([02Hb]) in the microenvironment of the tumor | 1 and 27 days
  Vascularization and perfusion enhance in the microenvironment of the tumor will be expressed as a relative increase of oxyhemoglobin concentration ([02Hb]) measured by functional near-infrared spectroscopy (fNIRS).
Relative deoxyhemoglobin concentration ([HHb]) in the microenvironment of the tumor | 1 and 27 days
  Vascularization and perfusion decrease in the microenvironment of the tumor will be expressed as a relative increase of deoxyhemoglobin concentration ([HHb]) measured by functional near-infrared spectroscopy (fNIRS).
Oxygen saturation (StO2) in the microenvironment of the tumor | 1 and 27 days
  Vascularization and perfusion enhance in the microenvironment of the tumor will be expressed as a relative increase of Oxygen saturation (StO2) measured by functional near-infrared spectroscopy (fNIRS).
Blood flow (BF) in the microenvironment of the tumor | 1 and 27 days
  Vascularization enhance in the microenvironment of the tumor will be expressed as a relative increase of blood flow index (BFI) measured by diffuse correlation optical spectroscopy (DCS).

SECONDARY OUTCOMES:
Height | 0, 28,and 35 days
  As complementary anthropometric measurement, we will include height measured in cm
Body mass | 0, 28,and 35 days
  As complementary anthropometric measurement, we will include body mass in kg.
Body mass index | 0, 28,and 35 days
  Body mass index will be calculated following the formula BMI=body mass / height^2.
Wait circumference | 0, 28,and 35 days
  As complementary anthropometric measurement, we will include waist circumference in cm.
Anthropometric measurements | 0, 28,and 35 days
  As complementary anthropometric measurement, we will include hip circumference in cm.
Bioimpedance measurements | 0, 28,and 35 days
  Water composition estimated by bioimpedance will be used to better estimate body composition
Maximal heart rate | 0, 28,and 35 days
  Maximal heart rate (HRmax) measured via a heart rate monitor synchronized with the gas analyzer during the incremental test.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Busquets, PhD, Principal Investigator — Institut Nacional d'Educació Física de Catalunya; Lucia Sagarra-Romero, PhD, Principal Investigator — Universidad San Jorge
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
After finishing the study, the data processed and anonymized will be available in B2share repositories (https://b2share.eudat.eu/) under the Creative Commons CC BY-NC-SA license.They will only be used for scientific purposes and after requesting permission from the authors and under the same conditions that we have established. The following data will not be made publicly available:
  * Personal data and other data that can be tracked to participants identity.
  * Data that compromises the protection of a partner(s) intellectual property.
  * The level of data made available will also be considered, for example, preprocessed data will not be provided unless there is a clear reason for doing so.
  * Datasets which cannot be shared because of legal and contractual reasons.
Supporting Information: Study Protocol, SAP
Time Frame: After finishing the study
Access Criteria: Once processing, quality control, organisation, analysis, and publication are complete, the data will be made accessible by deposition in open access repositories (https://b2share.eudat.eu).
  Members of the research team will form a data access committee. This committee will oversee that openly accessible data respect ethical and data security aspects, including intellectual property requirements. The possibilities of accessing the data in the specialized repository will always be decided in consultation with our collaborators.

REFERENCES:
- [Background] Chong F, Wang Y, Song M, Sun Q, Xie W, Song C. Sedentary behavior and risk of breast cancer: a dose-response meta-analysis from prospective studies. Breast Cancer. 2021 Jan;28(1):48-59. doi: 10.1007/s12282-020-01126-8. Epub 2020 Jun 30. PMID 32607943
- [Background] Lee K, Kruper L, Dieli-Conwright CM, Mortimer JE. The Impact of Obesity on Breast Cancer Diagnosis and Treatment. Curr Oncol Rep. 2019 Mar 27;21(5):41. doi: 10.1007/s11912-019-0787-1. PMID 30919143
- [Background] Gillis C, Loiselle SE, Fiore JF Jr, Awasthi R, Wykes L, Liberman AS, Stein B, Charlebois P, Carli F. Prehabilitation with Whey Protein Supplementation on Perioperative Functional Exercise Capacity in Patients Undergoing Colorectal Resection for Cancer: A Pilot Double-Blinded Randomized Placebo-Controlled Trial. J Acad Nutr Diet. 2016 May;116(5):802-12. doi: 10.1016/j.jand.2015.06.007. Epub 2015 Jul 21. PMID 26208743
- [Background] Santa Mina D, Hilton WJ, Matthew AG, Awasthi R, Bousquet-Dion G, Alibhai SMH, Au D, Fleshner NE, Finelli A, Clarke H, Aprikian A, Tanguay S, Carli F. Prehabilitation for radical prostatectomy: A multicentre randomized controlled trial. Surg Oncol. 2018 Jun;27(2):289-298. doi: 10.1016/j.suronc.2018.05.010. Epub 2018 May 7. PMID 29937184
- [Background] Sebio Garcia R, Yanez Brage MI, Gimenez Moolhuyzen E, Granger CL, Denehy L. Functional and postoperative outcomes after preoperative exercise training in patients with lung cancer: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):486-97. doi: 10.1093/icvts/ivw152. Epub 2016 May 25. PMID 27226400
- [Background] Bozzetti F. Forcing the vicious circle: sarcopenia increases toxicity, decreases response to chemotherapy and worsens with chemotherapy. Ann Oncol. 2017 Sep 1;28(9):2107-2118. doi: 10.1093/annonc/mdx271. PMID 28911059
- [Background] Lipsett A, Barrett S, Haruna F, Mustian K, O'Donovan A. The impact of exercise during adjuvant radiotherapy for breast cancer on fatigue and quality of life: A systematic review and meta-analysis. Breast. 2017 Apr;32:144-155. doi: 10.1016/j.breast.2017.02.002. Epub 2017 Feb 9. PMID 28189100
- [Background] Travier N, Velthuis MJ, Steins Bisschop CN, van den Buijs B, Monninkhof EM, Backx F, Los M, Erdkamp F, Bloemendal HJ, Rodenhuis C, de Roos MA, Verhaar M, ten Bokkel Huinink D, van der Wall E, Peeters PH, May AM. Effects of an 18-week exercise programme started early during breast cancer treatment: a randomised controlled trial. BMC Med. 2015 Jun 8;13:121. doi: 10.1186/s12916-015-0362-z. PMID 26050790
- [Background] Florez Bedoya CA, Cardoso ACF, Parker N, Ngo-Huang A, Petzel MQ, Kim MP, Fogelman D, Romero SG, Wang H, Park M, Katz MHG, Schadler KL. Exercise during preoperative therapy increases tumor vascularity in pancreatic tumor patients. Sci Rep. 2019 Sep 27;9(1):13966. doi: 10.1038/s41598-019-49582-3. PMID 31562341
- [Background] Ashcraft KA, Warner AB, Jones LW, Dewhirst MW. Exercise as Adjunct Therapy in Cancer. Semin Radiat Oncol. 2019 Jan;29(1):16-24. doi: 10.1016/j.semradonc.2018.10.001. PMID 30573180
- [Background] Schumacher O, Galvao DA, Taaffe DR, Chee R, Spry N, Newton RU. Exercise modulation of tumour perfusion and hypoxia to improve radiotherapy response in prostate cancer. Prostate Cancer Prostatic Dis. 2021 Mar;24(1):1-14. doi: 10.1038/s41391-020-0245-z. Epub 2020 Jul 6. PMID 32632128
- [Background] Betof AS, Lascola CD, Weitzel D, Landon C, Scarbrough PM, Devi GR, Palmer G, Jones LW, Dewhirst MW. Modulation of murine breast tumor vascularity, hypoxia and chemotherapeutic response by exercise. J Natl Cancer Inst. 2015 Mar 16;107(5):djv040. doi: 10.1093/jnci/djv040. Print 2015 May. PMID 25780062
- [Background] Jones LW, Viglianti BL, Tashjian JA, Kothadia SM, Keir ST, Freedland SJ, Potter MQ, Moon EJ, Schroeder T, Herndon JE 2nd, Dewhirst MW. Effect of aerobic exercise on tumor physiology in an animal model of human breast cancer. J Appl Physiol (1985). 2010 Feb;108(2):343-8. doi: 10.1152/japplphysiol.00424.2009. Epub 2009 Dec 3. PMID 19959769
- [Background] Durduran T, Choe R, Yu G, Zhou C, Tchou JC, Czerniecki BJ, Yodh AG. Diffuse optical measurement of blood flow in breast tumors. Opt Lett. 2005 Nov 1;30(21):2915-7. doi: 10.1364/ol.30.002915. PMID 16279468
- [Background] Nioka S, Chance B. NIR spectroscopic detection of breast cancer. Technol Cancer Res Treat. 2005 Oct;4(5):497-512. doi: 10.1177/153303460500400504. PMID 16173821
- [Background] Teng F, Cormier T, Sauer-Budge A, Chaudhury R, Pera V, Istfan R, Chargin D, Brookfield S, Ko NY, Roblyer DM. Wearable near-infrared optical probe for continuous monitoring during breast cancer neoadjuvant chemotherapy infusions. J Biomed Opt. 2017 Jan 1;22(1):14001. doi: 10.1117/1.JBO.22.1.014001. PMID 28114449
- [Background] Choe R, Durduran T. Diffuse Optical Monitoring of the Neoadjuvant Breast Cancer Therapy. IEEE J Sel Top Quantum Electron. 2012 Jul;18(4):1367-1386. doi: 10.1109/JSTQE.2011.2177963. Epub 2011 Dec 2. PMID 23243386
- [Background] Choe R, Putt ME, Carlile PM, Durduran T, Giammarco JM, Busch DR, Jung KW, Czerniecki BJ, Tchou J, Feldman MD, Mies C, Rosen MA, Schnall MD, DeMichele A, Yodh AG. Optically measured microvascular blood flow contrast of malignant breast tumors. PLoS One. 2014 Jun 26;9(6):e99683. doi: 10.1371/journal.pone.0099683. eCollection 2014. PMID 24967878
- [Background] Ramirez G, Proctor AR, Jung KW, Wu TT, Han S, Adams RR, Ren J, Byun DK, Madden KS, Brown EB, Foster TH, Farzam P, Durduran T, Choe R. Chemotherapeutic drug-specific alteration of microvascular blood flow in murine breast cancer as measured by diffuse correlation spectroscopy. Biomed Opt Express. 2016 Aug 24;7(9):3610-3630. doi: 10.1364/BOE.7.003610. eCollection 2016 Sep 1. PMID 27699124
- [Background] Rao R, Cruz V, Peng Y, Harker-Murray A, Haley BB, Zhao H, Xie XJ, Euhus D. Bootcamp during neoadjuvant chemotherapy for breast cancer: a randomized pilot trial. Breast Cancer (Auckl). 2012;6:39-46. doi: 10.4137/BCBCR.S9221. Epub 2012 Feb 1. PMID 22399859
- [Background] Busch DR, Choe R, Durduran T, Friedman DH, Baker WB, Maidment AD, Rosen MA, Schnall MD, Yodh AG. Blood flow reduction in breast tissue due to mammographic compression. Acad Radiol. 2014 Feb;21(2):151-61. doi: 10.1016/j.acra.2013.10.009. PMID 24439328
- [Background] Sagarra-Romero L, Butragueno J, Gomez-Bruton A, Lozano-Berges G, Vicente-Rodriguez G, Morales JS. Effects of an online home-based exercise intervention on breast cancer survivors during COVID-19 lockdown: a feasibility study. Support Care Cancer. 2022 Jul;30(7):6287-6297. doi: 10.1007/s00520-022-07069-4. Epub 2022 Apr 26. PMID 35471614
- [Background] Soriano-Maldonado A, Carrera-Ruiz A, Diez-Fernandez DM, Esteban-Simon A, Maldonado-Quesada M, Moreno-Poza N, Garcia-Martinez MDM, Alcaraz-Garcia C, Vazquez-Sousa R, Moreno-Martos H, Toro-de-Federico A, Hachem-Salas N, Artes-Rodriguez E, Rodriguez-Perez MA, Casimiro-Andujar AJ. Effects of a 12-week resistance and aerobic exercise program on muscular strength and quality of life in breast cancer survivors: Study protocol for the EFICAN randomized controlled trial. Medicine (Baltimore). 2019 Nov;98(44):e17625. doi: 10.1097/MD.0000000000017625. PMID 31689771
- [Background] Nahvijou A, Safari H, Yousefi M, Rajabi M, Arab-Zozani M, Ameri H. Mapping the cancer-specific FACT-B onto the generic SF-6Dv2. Breast Cancer. 2021 Jan;28(1):130-136. doi: 10.1007/s12282-020-01141-9. Epub 2020 Jul 25. PMID 32712768
- [Background] Klassen O, Schmidt ME, Scharhag-Rosenberger F, Sorkin M, Ulrich CM, Schneeweiss A, Potthoff K, Steindorf K, Wiskemann J. Cardiorespiratory fitness in breast cancer patients undergoing adjuvant therapy. Acta Oncol. 2014 Oct;53(10):1356-65. doi: 10.3109/0284186X.2014.899435. Epub 2014 May 16. PMID 24837860
- [Background] Morishita S, Wakasugi T, Tanaka T, Harada T, Kaida K, Ikegame K, Ogawa H, Domen K. Changes in Borg scale for resistance training and test of exercise tolerance in patients undergoing allogeneic hematopoietic stem cell transplantation. Support Care Cancer. 2018 Sep;26(9):3217-3223. doi: 10.1007/s00520-018-4168-3. Epub 2018 Apr 6. PMID 29626261
- [Background] Harrington S, Padua D, Battaglini C, Michener LA. Upper extremity strength and range of motion and their relationship to function in breast cancer survivors. Physiother Theory Pract. 2013 Oct;29(7):513-20. doi: 10.3109/09593985.2012.757683. Epub 2013 Jan 23. PMID 23343035
- [Background] Cortese L, Lo Presti G, Zanoletti M, Aranda G, Buttafava M, Contini D, Dalla Mora A, Dehghani H, Di Sieno L, de Fraguier S, Hanzu FA, Mora Porta M, Nguyen-Dinh A, Renna M, Rosinski B, Squarcia M, Tosi A, Weigel UM, Wojtkiewicz S, Durduran T. The LUCA device: a multi-modal platform combining diffuse optics and ultrasound imaging for thyroid cancer screening. Biomed Opt Express. 2021 May 14;12(6):3392-3409. doi: 10.1364/BOE.416561. eCollection 2021 Jun 1. PMID 34221667
- [Background] Cochran JM, Leproux A, Busch DR, O'Sullivan TD, Yang W, Mehta RS, Police AM, Tromberg BJ, Yodh AG. Breast cancer differential diagnosis using diffuse optical spectroscopic imaging and regression with z-score normalized data. J Biomed Opt. 2021 Feb;26(2):026004. doi: 10.1117/1.JBO.26.2.026004. PMID 33624457
- [Background] Zhou C, Choe R, Shah N, Durduran T, Yu G, Durkin A, Hsiang D, Mehta R, Butler J, Cerussi A, Tromberg BJ, Yodh AG. Diffuse optical monitoring of blood flow and oxygenation in human breast cancer during early stages of neoadjuvant chemotherapy. J Biomed Opt. 2007 Sep-Oct;12(5):051903. doi: 10.1117/1.2798595. PMID 17994886